CLINICAL TRIAL: NCT05216354
Title: An Open-Label, Phase 1 Study to Assess the Effect of Renal Impairment on the Pharmacokinetics of Fruquintinib
Brief Title: Fruquintinib Renal Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2021-013-00US2
Record Dates: First submitted 2022-01-19; First posted 2022-01-31 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (healthy subjects) (Experimental): 8 subject with normal renal function will be administered 5mg (1 x 5 mg capsule) fruquintinib
  Interventions: Drug: Fruquintinib
- Cohort 2 (severe renal impairment) (Experimental): 8 subjects with severe renal impairment will be administered 2 mg (2 x 1 mg capsules) fruquintinib
  Interventions: Drug: Fruquintinib
- Cohort 3 (moderate renal impairment) (Experimental): 8 subjects with moderate renal impairment will be administered 5 mg (a x 5 mg capsule) fruquintinib
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib will be administered as a single dose on the morning of Day 1 under fasting conditions
  Other Names: HMPL-013

SUMMARY:
A multicenter, open label, single-dose, single-period, sequential study to assess the effect of renal impairment on the pharmacokinetics of Fruquintinib

DETAILED DESCRIPTION:
This is a multicenter, open label, single-dose, single-period, sequential study in subjects without cancer with the primary objective of determining the effect of severe and moderate renal impairment on the PK of Fruquintinib. The secondary objective is to evaluate the safety in subjects severe and moderate renal impairment and subjects with normal function.

Initially, subjects with severe renal impairment and subjects with moderate renal impairment will be enrolled. Subjects with normal renal function will be enrolled after all other subjects have completed the study and will be matched for sex, age and body mass index. Subjects with renal impairment will be enrolled based on the renal function classification determined by Cockcroft-Gault scoring.

Subjects with severe renal impairment will receive a single dose of 2 mg fruquintinib to account for potential increase in fruquintinib pharmacokinetic (PK) exposure. Subjects with moderate renal impairment or normal renal function will receive a single dose of 5 mg fruquintinib.

ELIGIBILITY:
Inclusion Criteria:

All Subjects

* Male or female between the ages of 18 and 82 years old (inclusive)
* BMI >18 and ≤40 kg/m2 and body weight not <50 kg at screening.
* The subject is a non-smoker or light smoker who smokes no more than 10 cigarettes, 2 cigars, 2 pipes, or other nicotine equivalents (eg, vape, snuff, gum) of tobacco per day; willing to limit smoking during the treatment period to 4 cigarettes or 1 cigar per day.
* Females must be of non-childbearing potential or surgically sterile
* Males who have not had a successful vasectomy and are partners of women of childbearing potential must use, or their partners must use, a medically acceptable method of contraception starting for at least 1 menstrual cycle prior to and throughout the entire study treatment phase, and for 2 weeks after the last dose of study drug. Those with partners using hormonal contraceptives must also use an additional approved method of contraception such as a condom with spermicide. Males who have had a successful vasectomy (confirmed azoospermia, documentation needed) require no additional contraception.

Subjects with Renal Impairment

* For severe renal impairment, the subject must have CLcr of 15 to 29 mL/min at time of screening and day -1, as calculated by Cockcroft-Gault equation. For moderate renal impairment, the subject must have CLcr of 30 to 59 mL/min at time of screening and day -1, as calculated by Cockcroft-Gault equation. The difference between the screening and day -1 must be no more than 30%.
* The subject must have no clinically significant change in clinical condition within the last 30 days before screening, as documented by the subject's recent medical history.
* The subject must have a condition consistent with renal impairment and associated symptoms, but otherwise be determined to be in good health in the opinion of the Investigator.
* If diabetic, the subject must have the diabetes controlled (as determined by the Investigator).
* Concomitant medications to treat underlying disease states or medical conditions related to renal impairment are allowed. Subjects must be on a stable dose of medication and/or treatment regimen for at least 2 weeks before dosing as well as during the study.

Subjects with Normal Renal Function

* The subject must be without renal disease and have normal renal function
* The subject must be in good health

Exclusion Criteria:

All Subjects

* The subject has evidence of clinically significant cardiovascular, hepatic, GI, respiratory, endocrine, hematological, neurological, or psychiatric disease or abnormalities.
* The subject has a known history of any GI surgery or any condition possibly affecting drug absorption
* The subject has a clinically significant illness within 8 weeks or a clinically significant infection within 4 weeks prior to day 1.
* The subject has a clinically significant ECG abnormality.
* The subject has been diagnosed with acquired immune deficiency syndrome (AIDS), or tests positive for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
* The subject has participated in a clinical study of another drug before screening, and the time since the last use of other study drug is less than 5 times the half-life or 4 weeks before day 1, whichever is longer, or is currently enrolled in another clinical study.
* The subject has consumed grapefruit, starfruit, Seville oranges, or their products within 7 days prior to day 1.
* The subject has consumed herbal preparations/medications, including, but not limited to, kava, ephedra (ma huang), ginkgo biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng, within 7 days prior to day 1.
* The subject has received blood or blood products within 8 weeks, or donated blood or blood products within 8 weeks prior to day 1 or donated double red cells within 16 weeks prior to day 1.
* The subject has experienced a weight loss or gain of >10% within 4 weeks prior to day 1 as documented by recent medical history and weight at screening to check-in.
* The subject has used any drug that is a strong inhibitor or inducer of CYP3A within 2 weeks (within 3 weeks for St. John's Wort) prior to day 1 or will require use during the treatment period.
* The subject is allergic to the study drug or to any of its excipients.
* Female subject who is pregnant or planning to become pregnant, lactating, or breastfeeding.
* Male subject who plans to donate sperm or father a child within 3 months after receiving the study drug.
* The subject has any condition that would make them, in the opinion of the Investigator or Sponsor, unsuitable for the study, or who, in the opinion of the Investigator, is not likely to complete the study for any reason.

Subjects with Renal Impairment

* The subject has clinically significant vital sign abnormalities at screening or day -1.
* The subject has used acetaminophen at doses >1 g/day within 2 weeks prior to study drug administration.
* The subject has a history of drug or alcohol misuse within 6 months prior to screening or a positive drug test at screening or on day -1. A positive drug test may not be exclusionary if it is deemed to be the result of an approved prescribed concomitant medication.
* The subject has clinically significant, laboratory, or ECG findings (apart from those parameters that are related to impaired renal function or underlying disease [eg, diabetes, hypertension]) that, in the opinion of the Investigator, may interfere with any aspect of the study conduct or interpretation of the results.
* The subject has any history of renal transplant.
* The subject has any known significant bleeding diathesis (eg, history of recent bleeding from esophageal varices) that could preclude multiple venipuncture or deep intramuscular injections.
* The subject has acute or exacerbating renal disease, fluctuating or rapidly deteriorating renal function as indicated by widely varying or worsening of clinical and/or laboratory signs of renal impairment within 2 weeks of first dose.
* The subject has systolic blood pressure >180 mmHg or diastolic blood pressure >100 mmHg at screening or day -1

Subjects with Normal Renal Function

* The subject has evidence of clinically significant renal disease or abnormalities.
* The subject has evidence of a clinically significant deviation from normal in the physical examination, vital signs, or clinical laboratory determinations at screening or day -1
* The subject has a history of drug or alcohol misuse within 6 months prior to screening or a positive drug test at screening or day -1
* The subject has used any prescription or non-prescription drugs, including over-the-counter (OTC) medications or vitamins, within 2 weeks prior to day 1.
* The subject has systolic blood pressure >150 mmHg or diastolic blood pressure >95 mmHg at screening or day -1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
AUC 0-t | Day 1 to Day 11
  Area under the plasma concentration-time curve from time 0 to time of the last measurable concentration
AUC 0-inf | Day 1 to Day 11
  Area under the plasma concentration-time curve from time 0 to infinity (if data permit)
Maximum Plasma Concentration [Cmax] | Day 1 to Day 11
  To determine the maximum observed plasma concentration of Fruquintinib

SECONDARY OUTCOMES:
Incidence of AEs/SAEs | Day 1 to Day 11
  Any untoward medical occurrence associated with the use of study drug

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida